CLINICAL TRIAL: NCT02450175
Title: Etiology of the Platelet-Cancer Metastatic Pathway - A Study of Inflammatory Markers, Platelet Characteristics and Metastatic Surrogates in Cancer Patients and Controls
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinai Hospital of Baltimore (Other)
Responsible Party: Principal Investigator, Kenneth Miller, M.D., Medical Oncologist, Sinai Hospital of Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EOTPCMP
Record Dates: First submitted 2015-05-18; First posted 2015-05-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Neoplasm
Keywords: Platelet Activation; metastasis
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Everolimus; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cases (No Intervention): Patients with cancer whose platelets are examined
- Control (Placebo Comparator): Patients without cancer whose platelets are examined for comparison
  Interventions: Drug: Everolimus; Drug: Letrozole

INTERVENTIONS:
Drug: Everolimus — 10 mg of Everolimus daily (by mouth)
  Arms: Control
Drug: Letrozole — 2.5mg taken daily (by mouth)
  Arms: Control

SUMMARY:
The purpose of this research study is to understand if platelets in the blood become more active during cancer and specially advanced stages of cancer, in the future the investigators want to see if reducing platelet activity can improve survival in advanced cancer.

DETAILED DESCRIPTION:
Hypotheses for proposed study

Platelet reactivity as measured by percentage aggregation in response to agonists such as ADP is increased in patients with metastatic cancer compared to age sex and ethnicity matched controls.

Platelet activation as measured by release of cytokines and vasoactive substances such as VEGF, TGF-beta, and PDGF is increased in patients with metastatic cancer compared to age sex and ethnicity matched controls.

Study Design:

Single center matched case control design; matching variables are age, sex and ethnicity

Inclusion Criteria

Cases:

25 adult patients (>18 years old) with any form of metastatic or advanced stage (TNM stage III or equivalent) solid adenocarcinoma including breast, colon, and lung cancer will be eligible for inclusion in this study with no restrictions related to previous chemotherapy, radiotherapy, biological therapy or surgical management at the time of enrollment or in the past., although we will prefer to recruit them prior to initiating chemotherapy.

Controls:

25 patients will be selected based on age (+/- 5 years), sex and ethnicity matches from the outpatient medicine Clinic at Sinai hospital, as well as the Sinai community care clinic.

Exclusion Criteria:

Thrombocytopenia, defined as a platelet count of <100,000 at the time of recruitment of in the last available laboratory data

History of known bleeding disorder or known platelet dysfunction

Patients on antiplatelet treatment or anticoagulant therapies at the time of enrollment or 10 days prior to testing

CKD stage IV or greater

ELIGIBILITY:
Inclusion Criteria:

Cases:

25 adult patients (>18 years old) with any form of metastatic or advanced stage (TNM stage III or equivalent) solid adenocarcinoma including breast, colon, and lung cancer will be eligible for inclusion in this study with no restrictions related to previous chemotherapy, radiotherapy, biological therapy or surgical management at the time of enrollment or in the past., although we will prefer to recruit them prior to initiating chemotherapy.

Controls:

25 patients will be selected based on age (+/- 5 years), sex and ethnicity matches from the outpatient medicine Clinic at Sinai hospital, as well as the Sinai community care clinic.

Exclusion Criteria:

* Thrombocytopenia, defined as a platelet count of <100,000 at the time of
* recruitment of in the last available laboratory data
* History of known bleeding disorder or known platelet dysfunction
* Patients on antiplatelet treatment or anticoagulant therapies at the time of enrollment or 10 days prior to testing
* CKD stage IV or greater

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Platelet reactivity | 1 day

SECONDARY OUTCOMES:
Release of vasoactive substances, e.g. TGF Beta, | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- SInai Hospital of Baltimore, Inc., Baltimore, Maryland, United States